CLINICAL TRIAL: NCT00339339
Title: Bisphenol A and Metabolites in Urine and Saliva Associated With Placement of Composite Restorations
Brief Title: Levels of Bisphenol A in Urine and Saliva Following Placement of Composite Restorations
Status: Completed | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999904253; 04-D-N253
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2013-01-22

CONDITIONS: Dental Restorations
Keywords: Dental Materials; Resins; BisDMA; Absorption; Systemic

SUMMARY:
This study will determine whether placement of composite (white) dental restorations (fillings) increases concentrations of bisphenol A (BPA) and its metabolites in saliva and urine. These compounds have estrogenic-like properties that have raised concerns about their safety. Small amounts of the chemicals can leach out of dental sealants and be detected in saliva soon after the sealants are applied. Dental composites also contain some of these compounds.

U.S. Commissioned Corps officers who need fillings as part of their regular dental treatment and who select composite (white) restorations instead of amalgam (metal) may be included in this protocol. Participants are recruited from among officers receiving dental care at the commissioned officers dental clinic in Rockville, Md.

Participants complete a 15-minute interview to gather information about their recent diet and eating patterns. They also provide 3 to 4 urine and saliva samples, some collected before their dental restoration and some after treatment.

DETAILED DESCRIPTION:
A study by Olea et al in 1996 reported quantities of specific estrogenic compounds, Bisphenol A (BPA), bis-glycidyl methacrylate (bis-GMA) and Bis-A-dimethacrylate (bis-DMA) in saliva associated with the placement of certain dental sealants. This report raised concern regarding the safety of dental sealants and composite restorations. In a subsequent study bis-GMA was found to be stable, but bis-DMA was shown to hydrolyze to BPA, which likely accounts for the BPA detected in extracts from certain sealants. Another study reported detectable amounts of triethylene glycol dimethacrylate (TEGDMA) and BPA diglycidyl ether (BADGE) were released from sealants into saliva. All of these compounds have been shown to have deleterious effects for specific endpoints in vitro and various endocrine disruptive effects in some animal models, although results have not been consistent across animal strain, mode of administration, diet and other unknown factors. Detectable levels in plasma have not been shown.

Since there are insufficient data on the leachability concentrations in body fluids of these compounds associated with composite fillings in humans it is important to determine whether or not there are detectable levels of these compounds associated with the placement of composite restorations, and if so, whether the levels are sufficiently below the maximum acceptable or reference dose established by the EPA. For bisphenol A the maximum acceptable dose is 0.05 milligrams per kilogram of body weight per day (US EPA, 1993).

The National Institute of Dental and Craniofacial Research, the National Toxicology Program of the National Institute of Environmental Health Sciences, and the Commissioned Officers Dental Clinic Dentists have a unique opportunity to conduct a collaborative investigation at the Commissioned Officers Dental Clinic (CODC) in Rockville, MD involving commissioned officers who need dental restorations. This study will determine whether or not the placement of composite restorations is associated with the presence of these compounds in saliva. This is particularly timely since the number of composite restorations placed by dentists practicing in the U.S is rapidly increasing with over 80 million composite restorations placed in 1999 (ADA, 2001). It is of relevance to the U.S. Public Health Service Commissioned Officers Dental Clinic (CODC) because the CODC places composite materials in its dental clinic and wants to ensure that commissioned officers are receiving the best and safest possible dental care.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individual patients who require at least one restoration are eligible. We will give preference to patients who require multiple restorations that qualify for a composite filling material. Every attempt will be made to adequately represent women and minorities into the study.

EXCLUSION CRITERIA:

Individual patients who have received composite restorations or pit and fissure sealants during the past 3 months and individuals who wear removable dental appliances, such as orthodontic retainers or partial dentures, will be excluded.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 172 (Actual)
Dates: Start 2004-07-26; Study Completion 2013-01-22

CONTACTS AND LOCATIONS:
Overall Officials: Albert Kingman, Ph.D., Principal Investigator — National Institute of Dental and Craniofacial Research (NIDCR)
Locations (2):
- United States (2):
  - Commissioned Officers Dental Clinic (CODC), Rockville, Maryland
  - Kessler Air Force Base Dental Clinic, Biloxi, Mississippi

REFERENCES:
- [Derived] Kingman A, Hyman J, Masten SA, Jayaram B, Smith C, Eichmiller F, Arnold MC, Wong PA, Schaeffer JM, Solanki S, Dunn WJ. Bisphenol A and other compounds in human saliva and urine associated with the placement of composite restorations. J Am Dent Assoc. 2012 Dec;143(12):1292-302. doi: 10.14219/jada.archive.2012.0090. PMID 23204083